CLINICAL TRIAL: NCT04629898
Title: The Influence of Level of Immersion on Training Effects of Exergaming for Persons With Schizophrenia Spectrum Disorder
Brief Title: Level of Immersion of Virtual Reality and Cognition and Motor Performance in Patients of Schizophrenia Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Jen-Suh Chern, Associate Professor, National Taiwan Normal University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 201612HM014
Record Dates: First submitted 2020-11-06; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Schizophrenia; Virtual Reality; Video Games; Multi-tasks
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: multi-task in the real world and virtual reality video sport games — This was a 2-staged intervention study. The 1st stage intervention uses multitasks in the real world including stepping exercise, ball-kicking activity and bean-bag tossing activity. The 2nd stage intervention used video sport games conveyed by Xbox Kinect. Tennis and golf games were selected.

SUMMARY:
Schizophrenia Spectrum Disorder (SSD) is the main diagnosis in subjects with mental disability. The number of disabled SSD increased yearly and might be due to the ineffective medical and rehabilitative interventions on improving cognitive and motor function. Innovative and effective training programs are needed to decrease financial burden of medical care and social welfare.

Multi-tasks in real world were found to be effective in improving the sports skill of athletes and multi-tasking ability in the real world. No any study investigates in depth how the multi-tasks affect SSD patients' cognitive and motor performance.

Virtual reality exergaming (VREG) is a new form of multi-tasks incorporating information technology. It has been proved as an effective intervention media for patients with SSD in the single domain of physical fitness. No study exists examining its simultaneous influence in cognition and motor performance in SSD patients.

The purpose of this study is to examine the effects of different forms of multi-tasks on the cognitive and motor performance. The results of this study might be used by clinician treating patients with SSD in clinical decision making regarding to whether or not incorporating contemporary information technology in daily intervention and, furthermore, benefit the SSD more than using only the multi-task in the real world.

A total of 25 patients were recruited and participated in this study. They underwent 2-stage multi-task training. The first stage training used multi-tasks in the real world; the second stage training used new forms of multi-tasks which is virtual reality video sport games conveyed by Xbox Kinect. The training in each stage last for 12 weeks and there were 2 sessions in each week. The training duration in each session was 40 minutes.

All participants were measured at the following three time points: before any training begins, after the 1st stage of training and after the 2nd stage of training. The outcome measures include: upper limb motor function (measured by Box-and-Block Test), cognitive function (measured by Color Trail Test), functional mobility measured by Timed-Up-and-Go Test, and standing stability in 6 stance conditions, and voluntary center of gravity shifts during Functional Reach Test (measured by Footscan pressure measurement system).

ELIGIBILITY:
Inclusion Criteria:

* (1) diagnosed as schizophrenia or schizoaffective disorder by senior psychiatrists according to DSM-IV criteria and the disease onset was >1 year ago, (2) been judged as symptomatically stable by therapists, (3) was free of interfering or uncontrolled behaviors, (4) could stand independently for at least 3 minutes and walk 10 m without any mobility aids, (5) was ≥18 years old during recruitment for this study, (6) willing to participate in the study voluntarily

Exclusion Criteria:

* Patients were excluded if they were diagnosed with musculoskeletal impairment in the past year, had significant visual and auditory impairments, with severe cognitive impairment (based on Mini Mental State Examination score < 18), or were unable to follow verbal instructions or training and evaluation regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
The changes of Color Trail Test (CTT) | Measured at one week before and after the 1st stage training begin and one week after the end of the 2nd stage intervention
  There are two subtests: CTT1 & CTT2. The time spend to complete the two subtest is used representing executive function of the participants.
The changes of Box-and-Block Test | Measured at one week before and after the 1st stage training begin and one week after the end of the 2nd stage intervention
  This is a measure of upper limb motor performance. The number of blocks moved in one minute is the score of performance.Both the right and the left arm are tested.
The changes of Timed-Up-and-Go Test | Measured at one week before and after the 1st stage training begin and one week after the end of the 2nd stage intervention
  The time spend on completing the following task: standing up from a armless chair, walking ahead for 3 meteters, walking around a stool, walking back to the original chair and sitting down.
The changes of Postural sway while standing quietly | Measured at one week before and after the 1st stage training begin and one week after the end of the 2nd stage intervention
  The participants are instructed to stand on a 0.5 meter pressure measurement plate in 3 different standing posture (bilateral foot shoulder width apart, bilateral feet side by side, and tandem stance) and two visual conditions (eyes open v.s. closed. Coordinates of center of pressure(COP) are recorded and output and the the total path length of COP is calculated. The longer the COP path length, the poorer the postural stability.
The changes of Voluntary postural sway | Measured at one week before and after the 1st stage training begin and one week after the end of the 2nd stage intervention .
  The participants are instructed to stand on a 0.5 meter pressure measurement plate when performing the Functional Reach Test. Coordinates of center of pressure(COP) are recorded and output and the total path length of COP is calculated. The longer the COP path length, the better the dynamic postural control.

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Suh Chern, PhD, Principal Investigator — National Taiwan Normal University
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chien TY, Chern JS, Wang SP, Yang Y. Effects of multitask training on cognition and motor control in people with schizophrenia spectrum disorders. PLoS One. 2022 Jun 30;17(6):e0264745. doi: 10.1371/journal.pone.0264745. eCollection 2022. PMID 35771832